CLINICAL TRIAL: NCT00082810
Title: A Phase II Trial of Tipifarnib (R115777, Zarnestra™) in Combination With Fulvestrant (Faslodex®) in Postmenopausal Hormone Receptor-Positive Breast Cancer
Brief Title: Tipifarnib and Fulvestrant in Hormone Receptor-Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02982; 6205 (Other: CTEP); N01CM62204 (NIH)
Record Dates: First submitted 2004-05-14; First posted 2004-05-19 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Estrogen Receptor-positive Breast Cancer; Recurrent Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; tipifarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (tipifarnib, fulvestrant) (Experimental): Patients receive fulvestrant intramuscularly on day 1 and oral tipifarnib twice daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity*.
  Interventions: Drug: fulvestrant; Drug: tipifarnib

INTERVENTIONS:
Drug: fulvestrant — Given intramuscularly
  Other Names: Faslodex; ICI 182,780
Drug: tipifarnib — Given IV
  Other Names: R115777; Zarnestra

SUMMARY:
This phase II trial is studying how well giving tipifarnib together with fulvestrant works as second-line therapy in treating postmenopausal women with hormone receptor-positive inoperable locally advanced or metastatic breast cancer that has progressed after previous first-line endocrine therapy. Tipifarnib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using fulvestrant may fight breast cancer by blocking the use of estrogen. Combining tipifarnib with fulvestrant may kill tumor cells that did not respond to first-line therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of tipifarnib (R115777, Zarnestra™) in combination with fulvestrant based on clinical benefit rate (CBR, a combination of complete response rate, partial response rate, and stable disease for more than 24 weeks) in postmenopausal women with hormone receptor-positive metastatic breast cancer who have progressive disease after first-line endocrine therapy.

SECONDARY OBJECTIVES:

I. To determine the median time to progression (TTP) and duration of response of tipifarnib (R115777, Zarnestra™) in combination with fulvestrant in postmenopausal women with hormone receptor-positive metastatic breast cancer.

II. To determine the median overall survival of tipifarnib (R115777, Zarnestra™) in combination with fulvestrant in postmenopausal women with hormone receptor- positive metastatic breast cancer who have progressive disease after first-line endocrine therapy.

III. To determine the toxicity profile of tipifarnib (R115777, Zarnestra™) in combination with fulvestrant versus fulvestrant alone (from historical control) in postmenopausal women with hormone receptor positive metastatic breast cancer who have progressive disease after first-line endocrine therapy.

OUTLINE:

Patients receive fulvestrant intramuscularly on day 1 and oral tipifarnib twice daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity*.

NOTE: *Fulvestrant continues even if tipifarnib is held for toxicity.

Patients are followed every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed adenocarcinoma of the breast
* Patients must be postmenopausal
* Patients must have stage IV disease or inoperable locally advanced disease
* Patients must have ER- and/or PR-positive disease as determined by their local pathology laboratory
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan; all sites of disease should be noted and followed
* Prior hormonal therapy as adjuvant therapy and/or for metastatic disease is permitted; patients previously treated with two or more prior doses of fulvestrant are not eligible; patients who have received one prior dose of fulvestrant within 28 days are eligible so long as they meet other eligibility criteria
* Patients must have ECOG performance status 0-2 (Karnofsky >= 60%)
* Patients must have life expectancy of greater than 3 months
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin =< 2 mg/dL
* AST(SGOT)/ALT(SGPT) =< 2.5 x institutional upper limit of normal
* Creatinine less than or equal to 1.5 times the institutional upper limits of normal
* Patients must be disease-free of prior invasive malignancies for >= 5 years with the exception of: curatively-treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix
* Patients must have the ability to understand and the willingness to sign a written informed consent document
* Patients who have had previous therapy with farnesyltransferase inhibitor

Exclusion Criteria:

* Patients who have had radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier; patients who have had prior chemotherapy for metastatic disease are not eligible; prior adjuvant or neoadjuvant chemotherapy is allowed
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to tipifarnib (R115777, Zarnestra™) or other agents used in the study (e.g., imidazoles, quinolones)
* Presence of rapidly progressive, life-threatening metastases; this includes patients with extensive hepatic involvement (> 50% of the liver involved), symptomatic lymphangitic metastases, or brain or leptomeningeal involvement
* Concomitant anticancer treatment with the following exceptions: (1) bisphosphonates for bone metastases, (2) a GnRH analog is permitted if the patient had progressive disease on a GnRH analog plus a SERM or an AI; the GnRH analog may continue but the SERM or AI must be discontinued
* Grade 2 or more peripheral neuropathy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with tipifarnib or other agents administered during the study.; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2004-03; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Vahdat, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Li T, Christos PJ, Sparano JA, Hershman DL, Hoschander S, O'Brien K, Wright JJ, Vahdat LT. Phase II trial of the farnesyltransferase inhibitor tipifarnib plus fulvestrant in hormone receptor-positive metastatic breast cancer: New York Cancer Consortium Trial P6205. Ann Oncol. 2009 Apr;20(4):642-7. doi: 10.1093/annonc/mdn689. Epub 2009 Jan 19. PMID 19153124

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 33 patients were enrolled from 3 institutions between March 2004 and August 2006. Two patients were ineligible; one had a performance status of three and elevated liver function tests that exceeded inclusion criteria, whereas the other received prior chemotherapy for metatstatic disease.
Groups:
- Fulvestrant 250 mg + Tipifarnib 300 mg: Patients receive fulvestrant 250 mg intramuscularly on day 1 and oral tipifarnib 300 mg twice daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity
Period: Overall Study
Arm/Group | Fulvestrant 250 mg + Tipifarnib 300 mg
Started | 33
Completed | 2
Not Completed | 31
Not completed — Adverse Event | 3
Not completed — Progressive disease | 24
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Fulvestrant 250 mg + Tipifarnib 300 mg
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: years] | 61.0 [39 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Whites | 14
  Black | 3
  Hispanic | 14
  Asian | 2

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR) (CR Rate, PR Rate, and SD)
Description: Number of participants met the definition of Clinical Benefit Rate.Tumor response was assessed every three cycles by CT using RECIST (Response Evaluation Criteria In Solid Tumors) criteria. Per Response Evaluation Criteria in Solid Tumors (RECIST 1.0) for target lesions: Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD; Progressive Disease (PD): At least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter since the treatment started or the appearance of one or more new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Up to 24 weeks
Measure: Number; unit: participants
Arm/Group | Fulvestrant 250 mg + Tipifarnib 300 mg
Number analyzed (Participants) | 31
participants
  Partial response | 11
  Stable disease | 5
  Complete response | 0

2. Secondary Outcome: Time to Progression (TTP)
Description: TTP was estimated using the Kaplan-Meier method.
Time Frame: From randomization until progression of the disease, assessed up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fulvestrant 250 mg + Tipifarnib 300 mg
Number analyzed (Participants) | 31
months | 7.2 [2.8 to 9.8]

3. Secondary Outcome: Duration of Response
Description: DOR was defined for responders as the time from the onset of first response to disease progression and for non-responders as zero
Time Frame: Up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fulvestrant 250 mg + Tipifarnib 300 mg
Number analyzed (Participants) | 16
months | 16 [5.2 to 19.4]

4. Secondary Outcome: Toxicity as Assessed by NCI CTCAE Version 3.0
Description: Number of Participants with serious (grade 3) or life-threatening (grade 4) adverse events
Time Frame: Up to 4 years
Population: All treated patients who received at least one dose of tipifarnib were included in the safety analysis. A total of 342 cycles of therapy were administered (median 7 cycles/patient range 1-36 cycles)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Tipifarnib, Fulvestrant)
Number analyzed (Participants) | 33
Participants | 33

5. Secondary Outcome: Median Overall Survival
Description: The 95% confidence intervals will be used.
Time Frame: From randomization until death or censored at the date of last follow-up, assessed up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fulvestrant 250 mg + Tipifarnib 300 mg
Number analyzed (Participants) | 31
months | 19.4 [16.1 to 27.6]

ADVERSE EVENTS:
Arm/Group | Fulvestrant 250 mg + Tipifarnib 300 mg
Serious Adverse Events (participants affected / at risk) | 20/33
Other Adverse Events (participants affected / at risk) | 15/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant 250 mg + Tipifarnib 300 mg (N=33)
Neutropenia (Blood and lymphatic system disorders) | 4
Anemia (Blood and lymphatic system disorders) | 2
Infection (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 1
Cardiac Ischemia (Cardiac disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Insomnia (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 1
Ataxia (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine (Renal and urinary disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant 250 mg + Tipifarnib 300 mg (N=33)
Anemia (Blood and lymphatic system disorders) | 8
Infection (Infections and infestations) | 3
Nausea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 11
Anorexia (Metabolism and nutrition disorders) | 6
Fatigue (General disorders) | 12
Fever (General disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 5
Insomnia (Psychiatric disorders) | 4
Neuropathy (Nervous system disorders) | 7
Anxiety (Psychiatric disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Creatinine (Renal and urinary disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less